CLINICAL TRIAL: NCT02541097
Title: Preventing Language Decline in Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Regina Jokel, Clinician Associate, Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NPSASA-15-362999
Record Dates: First submitted 2015-08-31; First posted 2015-09-04 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Primary Progressive Aphasia
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Language Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Language therapy-Individual treatment (Active Comparator): Participants will receive intervention for naming impairment based on either phonological or semantic cues.
  Interventions: Behavioral: Language therapy
- Language therapy-Group treatment (Active Comparator): Following the individual therapy, participants will be randomly assigned to either verbal or non-verbal group
  Interventions: Behavioral: Language therapy

INTERVENTIONS:
Behavioral: Language therapy — Participants will receive semantic and phonological therapy for words they cannot retrieve spontaneously. They will be given an opportunity to practice the words in a group setting.

SUMMARY:
This study will establish factors fundamental to the improvement in communication and quality of life for people with dementia known as primary progressive aphasia (PPA). PPA is a type of dementia in which language declines but other cognitive skills (including memory) are preserved in the first several years after the onset. This makes those in the initial stages of PPA excellent candidates for treatment and creates a window of time (2-7 years) whereby they can lead independent lives with minimal support. However, currently, no communication therapy is available to people with PPA due to the progressive nature of the disorder and lack of awareness of available options for professionals willing to treat it.

Participants with PPA in our study will receive two kinds of therapy for the words they cannot recall spontaneously, and will be trained to maintain them through social interaction. The type of training will be based on the most successful interventions the investigators provided to people with PPA in our previous work. The investigators expect that successful re-learning of forgotten words and practicing them in a group setting will facilitate retention of communication skills leading to greater personal independence and increased/maintained quality of life for people with PPA. Our study represents natural combination of two novel approaches for PPA that ultimately will lead to lower demands on the health care system.

DETAILED DESCRIPTION:
The study will establish factors fundamental to the improvement in communication and quality of life for people with dementia known as primary progressive aphasia (PPA). PPA is a type of dementia in which language declines but other cognitive skills (including memory) are preserved in the first several years after the onset (see Mesulam 1982). This makes those in the initial stages of PPA excellent candidates for treatment and creates a window of time (2-7 years) whereby PPA individuals can lead independent lives with minimal support. However, currently, no communication therapy is available to people with PPA due to the progressive nature of the disorder and lack of awareness of available options for professionals willing to treat it.

Naming impairments are omnipresent in PPA. For this reason, anomia will be the focus of our intervention. Participants with PPA in our study will receive two kinds of therapy for the words they cannot recall spontaneously, and will be trained to maintain them through social interaction. The type of training will be based on the most successful interventions the investigators provided to people with PPA in our previous work (active encoding and errorless lerning). The investigators expect that successful re-learning of forgotten words and practicing them in a group setting will facilitate retention of communication skills leading to greater personal independence and increased/maintained quality of life for people with PPA. half of the cohort (randomly determined) will then participate in a communication group where conversations are encouraged and half will attend "non-verbal" group meetings when they will paint, watch movies and engage in other activities not requiring talking. To evaluate the benefits of practicing the re-learned words in a social setting naming skills will be tested for each participant before and after individual and group interventions.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of PPA
* fluent in English
* able to see and hear
* able to participate in individual and group sessions
* willing to travel to sessions
* physically independent (if assistive devices needed, must be able to operate them)

Exclusion Criteria:

* untreated mental conditions
* neurodegenerative conditions (other than PPA)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2018-12 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Naming accuracy measured with standard naming tests (e.g., BNT) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Regina Jokel, Principal Investigator — Rotman Research Institute, Baycrest and University of Toronto
Locations (1):
- Baycrest Health Sciences, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Only de-identified group data will be published